CLINICAL TRIAL: NCT06339554
Title: Alectinib-induced Endocrine Toxicity in Patients With ALK-positive Advanced NSCLC: an Onservational Study
Brief Title: Alectinib-induced Endocrine Toxicity
Acronym: TOSS-ALK
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Bria Emilio, Prof., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4806
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort A: Male ALK-positive ANSCLC patients receiving first-line treatment with alectinib
  Interventions: Drug: Alectinib 150 MG [Alecensa]
- Cohort B: Female ALK-positive ANSCLC patients receiving first-line treatment with alectinib
  Interventions: Drug: Alectinib 150 MG [Alecensa]
- Cohort C: Male ALK-negative ANSCLC patients receiving first-line treatment according to molecular profiling

INTERVENTIONS:
Drug: Alectinib 150 MG [Alecensa] — First line treatment for cohorts A and B
  Other Names: Alecensa
  Groups: Cohort A; Cohort B

SUMMARY:
The experimental Cohort A (male ALK+ ANSCLC patients receiving alectinib), the control Cohort B (female ALK+ ANSCLC patients receiving alectinib) and control Cohort C (male NON-ALK ANSCLC patients) were prospectively evaluated for full hormone assessment of androgen deficiency, AT 8 weeks after treatment start and in case of reported suspected symptoms. Patients with major sexual dysfunctions were referred to endocrinologist.

DETAILED DESCRIPTION:
Male patients (Cohorts A-C). After 8 weeks from treatment start (T1), as the same time of initial endocrine evaluation, we assessed symptoms of androgen deficiency by using the Androgen Deficiency in Aging Males (ADAM) questionnaire (Supplementary, SD1), a validated screening assessment of hypogonadism in adult males [15]. Next, the questionnaire was collected every 12 weeks during the routine clinic visits up to three years (if considered clinically appropriated). The response to the questionnaire was considered consistent with possible hypogonadism (i.e. positive), if the patient reported at least one major symptom (loss of libido and/or impotence; questions 1 and 7) or at least three minor symptoms. In case of suspected hypogonadism at ADAM questionnaire, hormonal tests were again performed and the patient was referred to Andrology Unit of the Endocrinology Departement in case of abnormal results. Andrology visit included physical examination, testicular and scrotum ultrasound, medical history and hormonal tests reviewing; when testosterone replacement and/or drugs for erectile dysfunction were prescribed, the overall effectiveness on symptoms of hypogonadism (improved/not improved) was assessed by the andrologist and checked at next oncologic visits.

Female patients (Cohort B). After 8 weeks from treatment start (T1), as the same time of initial endocrine assessment, we assessed symptoms of sexual dysfunctions, according to menopausal status, by using the EORTC QLQ - BR23 and FACT-B (Version 4) questionnaires. In case of clinically significant gynaecological symptoms and/or abnormal results of sexual hormones axis in relation to menopausal status, the patients were referred to multidisciplinary evaluation by an endocrinologist and a gynaecologist. Multidisciplinary evaluation included physical and gynaecological examination, pelvic ultrasound, medical history and hormonal tests reviewing; diagnosis and treatment of endocrine/gynaecological dysfunction and prescribed treatment/intervention were reported in medical history and checked at next oncologic visits

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced NSCLC (ANSCLC) For ALK+ NSCLC (Cohorts A-B) 1a. ALK-rearrangement confirmed by NGS and/or VENTANA ALK (D5F3) immunoistochemical assay 1b. Treatment naïve patients candidate to treatment with alectinib oral at standard dose of 600 mg twice daily
2. Patient aged 18 to 70 years
3. To be sexually active at time of enrolment
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
5. Written informed consent

Exclusion Criteria:

1. History of endocrine disorders, excepting for controlled hypothyroidism (surgical or non-surgical) treated with replacement levothyroxine since at least 2 years
2. Any cancer-related or medical condition that would interfere with the patient reported outcomes or laboratory assessment. Examples include, but are not limited to:

2a. Cancer-related conditions that may preclude/undermine sexual activity (e.g. leptomeningeal carcinomatosis, pathological vertebral fractures, gonadic metastases, unstable spinal cord compression, uncontrolled neurological symptoms, surgical complications)

2b. History of chronic liver disease or hormonal replacement therapy (e.g. ADT for prostatic cancer)

2c. Participants who not adequately recovered from previous confirmed chemotherapy-induced gonadotoxicity (e.g. cisplatin)

2d. Chronic use of drugs with known effect on male sexuality, including opiates, anxiolytics, antidepressants, mood stabilizers, beta blockers (e.g. atenolol) and high dose diuretics

2e. Psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study

2f. Major psychological disorder and/or high distress level that would interfere with sexual function and the participant's ability to cooperate with the requirements of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cohort A + C = male Cohort B = female
Study Population: TOSS-ALK is single-Institution observational prospective sex-based trial aimed to assess endocrine toxicity in ALK+ advanced/metastatic ANSCLC male patients treated with first-line alectinib (Cohort A). As control cohorts, we included female ALK+ ANSCLC patients (Cohort B) and male patients with NON-ALK+ NSCLC who are receiving active treatment (ACT) according to tumour molecular profiling (Cohort C).
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of endocrine toxicity in overall ALK-positive | Time from treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Percentege of endocrine alterations among patients included in Cohort A and B
Incidence of symptomatic hypogonadism in male ANSCLC patients | Time from treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Percentage of endocrine alterations and/or clinical sexual dysfuctions among male patients included in Cohort A and C

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, Italy